CLINICAL TRIAL: NCT04990063
Title: A Clinical Study on the Safety and Efficacy of Adoptive TKC Transfer Combined With Chemotherapy for Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Adoptive TKC Transfer Combined With Chemotherapy for Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: suhaichuan (Other)
Collaborators: Shanghai Biomed-union Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, suhaichuan, Associate Chief Physician, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHKYSW-TKC-CAN-102
Record Dates: First submitted 2021-07-16; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Advanced Non-small Cell Lung Cancer; Chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adoptive TKC transfer combined with chemotherapy (Experimental): NK cells and γδT cells are isolated from the patients' PBMCs obtained before standard chemotherapy and then co-cultured ex-vivo. Patients will receive multiple TKC treatments under administration, 3 weeks/cycle. The first infusion will be conducted in 7-10 days after chemotherapy and is assessed by the investigators. TKC cells are transfused to patients in a dosage escalated manner. Dose escalation starts at 1×10^8 cells/kg (based on the whole body weight). After the safety assurance of the initial administration, the next course, up to 8 courses, is resumed and the dose maybe increased subsequently at the discretion of the investigators, or reduced for safety reason.
  Interventions: Drug: Chemotherapy; Biological: Adoptive TKC transfer therapy

INTERVENTIONS:
Drug: Chemotherapy — Standard chemotherapy drug
Biological: Adoptive TKC transfer therapy — TKC: co-cultured autologous NK cells and γδT cells

SUMMARY:
Innate immune cells are an important part of the body's innate immune system, the first line of defense against infection and cancer. Tumor killer cells (TKC) are mixed cultures of two kinds of innate immune cells, namely natural killer cells (NK cells) and gamma delta T cells (γδT cells), which are co-activated and co-cultured ex-vivo in a certain proportion by the unique TKC technology. Adoptive TKC transfer is expected to exert a strong anti-tumor effect through synergistic action between NK cells and γδT cells. In this study, the safety, tolerance, and preliminary efficacy of adoptive TKC transfer combined with chemotherapy will be examined in patients with advanced NSCLC.

DETAILED DESCRIPTION:
Primary Objective:

● To describe the safety profile and toxicity tolerance of combining adoptive TKC transfer with chemotherapy in patients with advanced non-small cell lung cancer (NSCLC).

Secondary Objectives:

● To evaluate the preliminary efficacy of combining adoptive TKC transfer with chemotherapy in the treatment of advanced NSCLC.

Design:

* This is a single-centre, open label, non-randomised, no control clinical trial.
* NK cells and γδT cells are isolated from the patients' peripheral blood mononuclear cells (PBMCs) obtained before chemotherapy and then co-cultured with TKC technology ex-vivo. The mixed cultures will be used in multiple infusions under administration. The first infusion will be conducted in 7-10 days after chemotherapy and is assessed by the investigators.
* Clinical responses will be evaluated closely in about 30 days and last up to 2 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years old and ≤70 years old when signing the informed consent; regardless of gender;
2. Body weight>40kg;
3. Histopathology or cytology confirmed as advanced NSCLC which is not suitable for radical surgical resection;
4. At least one measurable lesion according to the RECIST 1.1 criteria; according to the CT or MRI cross-sectional imaging, the diameter of a single lesion ≤8 cm, or the maximum diameter of a single lesion ≤5 cm and the number of lesions ≤5 (including metastatic lesions).
5. Imaging examination showed no tumor thrombus in the portal vein/inferior vena cava;
6. Acceptable hemopoietic ability: hemoglobin (HGB) >90g/L (no blood transfusion within two weeks), absolute neutrophil count (ANC) >1.5×10^9/L, platelet count >1.0×10^11/L, absolute lymphocyte count (ALC)>500×10^9/L;
7. Prothrombin time (PT)/international normalized ratio (INR) <1.5 ULN and partial thromboplastin time (PTT)/activated partial thromboplastin time (APTT) <1.5 ULN;
8. Acceptable liver and kidney functions: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 ULN in subjects without liver metastases and ≤3.5 upper limit of normal (ULN) in those with liver metastases; bilirubin≤1.5 ULN (excluding hyperbilirubinemia or non-liver-derived hyperbilirubinemia); creatinine ≤1.5 ULN and creatinine clearance rate≥40 mL/min;
9. Women of child-bearing age must be negative for pregnancy test at 7 days before initiation of the treatment.
10. Eastern Cooperative Oncology Group (ECOG) scores≤1.
11. Expected survival no less than 6 months.

Exclusion Criteria:

1. History of any chemotherapy within 2 weeks before a single blood collection;
2. Participating in other clinical trials in the past 30 days;
3. Current on systemic steroid or steroid inhalers;
4. Active brain metastasis or spinal cord compression
5. Uncontrollable pleural and peritoneal effusion requiring clinical treatment or intervention;
6. Active bleeding, and thrombotic diseases requiring treatment;
7. Uncontrolled infectious diseases, such as baseline hepatitis B virus (HBV) DNA≥2000 IU/mL, positive for anti-human immunodeficiency virus （HIV） antibody and hepatitis C virus (HCV)-RNA; Other active infection with clinical significance;
8. Organ failure; Heart: Grade III and IV ; or with hypertension uncontrolled by the standard treatment, history of myocarditis or myocardial infarction within 1 year; Liver: Class C according to the Child-Turcottei-Pugh System (CTP); Kidneys: Kidney failure and uremic syndrome; Lungs: Serious symptoms of respiratory failure; Brain: Disturbance of consciousness;
9. Allergic diathesis and allergic to immunotherapy or relevant drugs;
10. Pregnancy or lactation;
11. History of other active malignancies in the past 5 years, excluding basal or squamous skin carcinoma, superficial bladder cancer, and breast cancer in situ which have completely healed and require no follow-up treatment;
12. Serious autoimmune diseases or immunodeficiency disease, including those with confirmed severe autoimmune diseases and requiring long-term use (over 2 months) of systemic immunosuppressants (steroids) or having immune-mediated symptomatic diseases, such as ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE) and autoimmune vasculitis (eg., Wegener's granulomatosis);
13. Any mental diseases, including dementia and changes in mental status that may influence the understanding about the informed consent and questionnaire;
14. Judged as serious uncontrollable diseases by the researchers, or other conditions that may interfere with the treatment and therefore being ineligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-08 (Estimated); Primary Completion 2022-08-08 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation by the incidence of adverse events (AEs) and serious adverse events (SAEs) | 24 months
  Incidence of AEs and SAEs of each participant will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate (ORR) | 24 months
  ORR is defined as the percentage of patients who have a clinical response (objective tumor regression).ORR is computed by: the sum of the number of patients with Complete Response (CR) and number of patients with Partial Response (PR) / total number of patients. The total number of patients is the sum of the number of patients with CR, PR, stable disease (SD) or progressive disease (PD). The Response Evaluation Criteria in Solid Tumors (RECIST v1.1) is used as the criteria to determine whether a tumor disappears (CR), shrinks (PR), stays the same (SD) or gets bigger (PD).
Duration of response (DOR) | 24 months
  DOR is the time between the initial response to treatment per RECIST v1.1 and subsequent disease progression among patients achieving Complete Response (CR) or Partial Response (PR). RECIST v1.1 is used as the criteria to determine whether a tumor disappears (CR) or shrinks (PR).
Progression-free survival (PFS) | 24 months
  PFS is the length of time from the date patient enrolled in to the date on which tumor progresses or the patient dies for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Helong Zhang, Study Chair — IEC of Institution for National Drug Clinical Trials ,Tangdu Hospital
Locations (1):
- Tangdu Hospital, Fourth Military Medical University, Xi’an, Shanxi, China